CLINICAL TRIAL: NCT02169440
Title: Effect of BIA 9-1067 on the Pharmacokinetics and Pharmacodynamics of Warfarin in Healthy Volunteers
Brief Title: Effect of BIA 9-1067 on the Pharmacokinetics and Pharmacodynamics of Warfarin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-116
Record Dates: First submitted 2012-01-24; First posted 2014-06-23 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-11

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson's disease (PD); BIA 9-1067; Opicapone
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Period 1: BIA 9-1067 + warfarin Period 2: warfarin
  Interventions: Drug: BIA 9-1067; Drug: Warfarin
- Group 2 (Active Comparator): Period 1: warfarin Period 2: BIA 9-1067 + warfarin
  Interventions: Drug: BIA 9-1067; Drug: Warfarin

INTERVENTIONS:
Drug: BIA 9-1067 — BIA 9-1067 25 mg
  Other Names: OPC, Opicapone
Drug: Warfarin — Warfarin 25 mg
  Other Names: Varfine®

SUMMARY:
The purpose of this study is to investigate CYP2C9 inhibition by BIA 9-1067 through the assessment of its effect on the pharmacokinetics of S-warfarin, a substrate of CYP2C9.

DETAILED DESCRIPTION:
Single-centre, open-label, randomised, two-way crossover study in healthy young male and female volunteers. The study was to consist of 2 treatment periods separated by a washout period of 14 days or more. In one period, subjects were to receive a single-dose of 25 mg BIA 9-1067 with a single-dose of racemic 25 mg warfarin. In the other period, a 25 mg warfarin single-dose was to be administered alone.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent.
* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* Healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Negative tests for HBsAg, anti-HCVAb and HIV-1 and HIV-2 Ab at screening.
* Clinical laboratory test results clinically acceptable at screening and admission to each treatment period.
* Negative screen for alcohol and drugs of abuse at screening and admission to each treatment period.
* Non-smokers or ex-smokers for at least 3 months.
* (If female) She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: double barrier or intrauterine device.
* (If female) She had a negative urine pregnancy test at screening and admission to each treatment period.

Exclusion Criteria:

* Clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Clinically relevant surgical history.
* Personal or family history of haemostatic disorder.
* Personal or family history of bleeding complications after surgery or tooth extraction, nose or gingival bleeding, or haemorrhagic diathesis.
* Any abnormality in the coagulation tests.
* Any abnormality in the liver function tests.
* A history of relevant atopy or drug hypersensitivity.
* History of alcoholism or drug abuse.
* Consumed more than 14 units of alcohol a week.
* Significant infection or known inflammatory process at screening or admission to each treatment period.
* Acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to each treatment period.
* Had used medicines within 2 weeks of admission to first period that may have affected the safety or other study assessments, in the investigator's opinion.
* Had previously received BIA 9-1067.
* Had used any investigational drug or participated in any clinical trial within 6 months prior to screening.
* Had participated in more than 2 clinical trials within the 12 months prior to screening.
* Had donated or received any blood or blood products within the 3 months prior to screening.
* Vegetarians, vegans or had medical dietary restrictions.
* Cannot communicate reliably with the investigator.
* Unlikely to co-operate with the requirements of the study.
* Unwilling or unable to gave written informed consent.
* Employees at BIAL - Portela & Co, SA.
* (If female) She was pregnant or breast-feeding.
* (If female) She was of childbearing potential and she did not used an approved effective contraceptive method (double-barrier or intra-uterine device) or she used oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- BIAL - Portela & Cª - Human Pharmacology Unit (UFH), S. Mamede Do Coronado, Trofa, Portugal

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: BIA 9-1067 + Warfarin, Then Warfarin: Period 1: BIA 9-1067 + warfarin Period 2: warfarin
  BIA 9-1067: BIA 9-1067 25 mg
  Warfarin: Warfarin 25 mg
- Group 2: Warfarin, Then BIA 9-1067 + Warfarin: Period 1: warfarin Period 2: BIA 9-1067 + warfarin
  BIA 9-1067: BIA 9-1067 25 mg
  Warfarin: Warfarin 25 mg
Period: Overall Study
Arm/Group | Group 1: BIA 9-1067 + Warfarin, Then Warfarin | Group 2: Warfarin, Then BIA 9-1067 + Warfarin
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: BIA 9-1067 + Warfarin, Then Warfarin | Group 2: Warfarin, Then BIA 9-1067 + Warfarin | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Plasma Concentration (BIA 9-1067 + Warfarin)
Description: Mean plasma BIA 9-1067 pharmacokinetic parameters obtained following an oral single dose of 25 mg warfarin co-administered with 25 mg BIA 9-1067
Time Frame: before dose and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 h post- dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- BIA 9-1067 + Warfarin: BIA 9-1067 25 mg + Warfarin 25 mg
Arm/Group | BIA 9-1067 + Warfarin
Number analyzed (Participants) | 20
ng/mL | 196 (106)

2. Primary Outcome: Tmax - Time to Maximum Observed Plasma Concentration (BIA 9-1067 + Warfarin)
Description: as for outcome 1
Time Frame: before dose and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 h post- dose.
Measure: Median (Full Range); unit: hours
Arm/Group | BIA 9-1067 + Warfarin
Number analyzed (Participants) | 20
hours | 3.00 [1.0 to 6.0]

3. Primary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve From Time 0 to Last Observed Concentration (BIA 9-1067 + Warfarin)
Description: as for outcome 1
Time Frame: before dose and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 h post- dose.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | BIA 9-1067 + Warfarin
Number analyzed (Participants) | 20
ng.h/mL | 610 (420)

4. Primary Outcome: Cmax = Maximum Plasma Concentration (Warfarin Alone)
Description: Mean plasma S-warfarin pharmacokinetic parameters obtained following an oral singledose of 25 mg warfarin administered alone
Time Frame: before dose and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 h post- dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Warfarin Alone: Warfarin 25 mg
Arm/Group | Warfarin Alone
Number analyzed (Participants) | 20
ng/mL | 1940 (364)

5. Primary Outcome: Tmax - Time to Maximum Observed Plasma Concentration (Warfarin Alone)
Description: as for outcome 4
Time Frame: before dose and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 h post- dose.
Measure: Median (Full Range); unit: hours
Arm/Group | Warfarin Alone
Number analyzed (Participants) | 20
hours | 2.50 [0.5 to 16.0]

6. Primary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve From Time 0 to Last Observed Concentration (Warfarin Alone)
Description: as for outcome 4
Time Frame: before dose and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 h post- dose.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Warfarin Alone
Number analyzed (Participants) | 20
ng.h/mL | 75098 (13792)

7. Primary Outcome: Cmax - Maximum Observed Plasma Concentration (Warfarin + BIA 9-1067)
Description: Mean plasma S-warfarin pharmacokinetic parameters obtained following an oral single dose of 25 mg warfarin co-administered with 25 mg BIA 9-1067
Time Frame: before dose and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 h post- dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Warfarin + BIA 9-1067: 25 mg warfarin + 25 mg BIA 9-1067
Arm/Group | Warfarin + BIA 9-1067
Number analyzed (Participants) | 20
ng/mL | 2003 (392)

8. Primary Outcome: Tmax - Time to Maximum Observed Plasma Concentration (Warfarin + BIA 9-1067)
Description: as for outcome 7
Time Frame: before dose and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 h post- dose.
Measure: Median (Full Range); unit: hours
Arm/Group | Warfarin + BIA 9-1067
Number analyzed (Participants) | 20
hours | 3.00 [0.5 to 8.0]

9. Primary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve From Time 0 to Last Observed Concentration (Warfarin + BIA 9-1067)
Description: as for outcome 7
Time Frame: before dose and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 h post- dose.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Warfarin + BIA 9-1067
Number analyzed (Participants) | 20
ng.h/mL | 78177 (15196)

ADVERSE EVENTS:
Groups:
- BIA 9-1067 + Warfarin: BIA 9-1067 25 mg Warfarin 25 mg
Arm/Group | BIA 9-1067 + Warfarin | Warfarin
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 6/20 | 7/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 9-1067 + Warfarin (N=20) | Warfarin (N=20)
Blepharitis (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Vessel puncture site haematoma (Injury, poisoning and procedural complications) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes